CLINICAL TRIAL: NCT02127372
Title: A Phase I - II Open Label Study of the Maximum Tolerated Dose, Safety and Efficacy of Docetaxel and Cisplatin Plus STI571 in Advanced Non-Small Cell Lung Cancer
Brief Title: Maximum Tolerated Dose, Safety and Efficacy of Docetaxel / Cisplatin + STI571
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was closed due to poor accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008205
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel; Cisplatin; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Docetaxel, Cisplatin and STI571 — Treatment will consist of docetaxel plus cisplatin IV every 21days and oral STI571 given on Days -5 to 2 with each chemotherapy cycle. A maximum of 6 cycles will be given.
  Phase 1 dose levels are:
  * Level 1 Docetaxel/Cisplatin 60 mg/m2, STI571 300mg
  * Level 2 Docetaxel/Cisplatin 60 mg/m2, STI571 400mg
  * Level 3 Docetaxel/Cisplatin 70 mg/m2, STI571 400mg
  * Level 4 Docetaxel/Cisplatin 70 mg/m2, STI571 600mg
  * Level 5 Docetaxel/Cisplatin 75 mg/m2, STI571 600mg
  * Level 6 Docetaxel/Cisplatin 75 mg/m2, STI571 800mg
  Once the MTD level has been established, the previous dose level will be the dosing schedule for Phase II.
  Other Names: Taxotere; Platinol; Gleevec; Imatinib
Drug: Docetaxel
  Other Names: Taxotere
Drug: Cisplatin
  Other Names: Platinol

SUMMARY:
This is a Phase 1/Phase 2 study of STI571 combined with docetaxel and cisplatin for treatment of patients with recurrent and metastatic Non-Small Cell Lung Cancer (NSCLC).

This research study has 2 parts to it. The first part (Phase 1) is called a dose-escalation. Not all subjects enrolled into this phase of the study will receive the same dose. The purpose of the dose-escalation is to determine the highest safe dose of STI571 that can be used in combination with docetaxel and cisplatin. That dose will be used in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically recurrent, or advanced NSCLC: Stage IV disease; or Stage IIIB due to malignant pleural effusion is allowed- only if successfully pleurodesed.
* Tumor tissue slides must express phosophorylated pdgf-rB by IHC.
* At least one measurable target lesion as defined by RECIST criteria that has not been irradiated.
* No prior chemotherapy treatment for this disease will be allowed. Patients with brain metastasis will have to be, after appropriate treatment, neurologically stable for at least 1-2 weeks (off steroids) prior to study enrollment.
* ECOG performance status 0-1.
* Meets initial laboratory parameters.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria

* Any prior treatment with a biologic response modifier or chemotherapeutic agent for this disease.
* Any concomitant malignancy except non-melanoma skin cancer or in-situ carcinoma of the cervix.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to STI571 and/or docetaxel, or other drugs formulated with polysorbate 80 and/or cisplatin.
* Patients with:

  * Contrast allergy.
  * GI bleed ≤ 1 month from study enrollment.
  * Intermittent or chronic oxygen requirements.
  * Pulse oximetry <90%.
  * Grade 3 dyspnea.
  * History of poorly regulated anticoagulation with warfarin.
  * Edema or fluid retention grade >1.
  * Neuropathy grade ≥1.
* Uncontrolled inter-current medical illness including, but not limited to, ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure, unstable angina pectoris, ≤3 months myocardial infarction or cardiac arrhythmia.
* Psychiatric illness/social situations that would limit compliance with study requirement or that would prevent informed consent or psychiatric illness/social situations requiring inpatient treatment within the past 3 months.
* Any type of hearing impairment.
* Known HIV infection.
* Receiving other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-11; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Vlahovic, MD, MHS, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Advanced Non-Small Cell Lung Cancer were enrolled from November 2004 to April 2009. The study was closed due to poor accrual.
Pre-assignment Details: Overall, 72 subject signed a consent form and 43 went on to start treatment on study.
  Of the 24 subjects who signed a consent form for Phase 1, 9 were screen failures and did not start study treatment.
  Of the 48 subjects who signed a consent form for Phase 2, 20 were screen failures and did not start study treatment.
Groups:
- Phase 1: Eligible subjects will be enrolled in the Phase I portion of the study to determine the MTD of STI571 in combination with docetaxel plus cisplatin, given every three weeks. STI will be given intermittently for 7 days (Day -5 to Day 2) When MTD is established, Phase II study will evaluate for combined modality safety, tolerability and efficacy (response rate vs. historical control). All subjects will start with STI571 therapy alone for 7 days; pre and post STI571 treatment (Days -8 and 0)
- Phase 2: The objective of this two-stage Phase II study is to determine whether the combination of STI571, docetaxel, and cisplatin merits inclusion in a randomized study for chemotherapy-naïve patients with advanced NSCLC. The dose for the Phase 2 portion of the trial will be IV Docetaxel / Cisplatin 60 / 60 mg/m2 and 400 mg STI571 PO QD
Period: Overall Study
Arm/Group | Phase 1 | Phase 2
Started | 15 (Signed Consent) | 28 (Signed Consent)
Started Study Treatment | 15 | 28
Completed | 14 (Completed at least one cycle and were available for dose limiting toxicity (DLT) evaluation.) | 28
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who started study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 15 | 28 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (12.5) | 60.0 (9.5) | 57.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 10 | 17 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 28 | 43

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) of STI571
Description: To determine the maximum tolerated dose (MTD) of STI571, docetaxel, and cisplatin, when administered in combination for the treatment of patients with chemo-naïve recurrent and metastatic (stage IV) NSCLC.
Time Frame: After cycle 1, day 22
Population: One patient only received the lead-in dose of STI571 prior to withdrawing from the study without a DLT. This subject is not included in the DLT determination.
Measure: Number; unit: mg
Arm/Group | Phase 1
Number analyzed (Participants) | 14
mg | 400

2. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) of Docetaxel and Cisplatin
Description: To determine the maximum tolerated dose (MTD) of STI571, docetaxel, and cisplatin when administered in combination for the treatment of patients with chemo-naïve recurrent and metastatic (stage IV) NSCLC.
Time Frame: After cycle 1, day 22
Population: as for outcome 1
Measure: Number; unit: mg/m2
Arm/Group | Phase 1
Number analyzed (Participants) | 14
mg/m2
  Docetaxel | 60
  Cisplatin | 60

3. Secondary Outcome: Phase 2: 1 Year Survival
Description: Phase II: Percentage of patients alive 1 year from the start of protocol treatment.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 28
percentage of participants | 61 [40 to 76]

4. Secondary Outcome: Change in Gd-MRI Measurement
Description: The change in Gd-MRI perfusion/permeability measurement between pre and post 7-day of STI571 treatment.
Time Frame: Day 7
Population: Because the study was terminated prior to completion, correlative studies were not run.
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Phase II - Radiographic Response
Description: The percentage of patients with a complete or partial response.
  Responses for the Phase II portion of the trial will be by Response Evaluation Criteria In Solid Tumors (RECIST) criteria as follows:
  Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: After Cycle 6, approximately 18 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 28
percentage of participants | 25 [11 to 45]

ADVERSE EVENTS:
Arm/Group | Phase 1 | Phase 2
Serious Adverse Events (participants affected / at risk) | 9/15 | 15/28
Other Adverse Events (participants affected / at risk) | 15/15 | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=15) | Phase 2 (N=28)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Stomach pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Edema face (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 3
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=15) | Phase 2 (N=28)
Anemia (Blood and lymphatic system disorders) | 7 | 17
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Blurred vision (Eye disorders) | 1 | 4
Dry eye (Eye disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 0 | 2
Flashing lights (Eye disorders) | 1 | 1
Watering eyes (Eye disorders) | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 8 | 6
Diarrhea (Gastrointestinal disorders) | 6 | 10
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 5
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 13 | 13
Vomiting (Gastrointestinal disorders) | 6 | 8
Chills (General disorders) | 1 | 1
Edema face (General disorders) | 3 | 2
Edema limbs (General disorders) | 5 | 10
Edema trunk (General disorders) | 1 | 1
Fatigue (General disorders) | 11 | 18
Fever (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 2 | 3
Allergic reaction (Immune system disorders) | 0 | 2
Gum infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Alkaline phosphatase increased (Investigations) | 0 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 2
Creatinine increased (Investigations) | 1 | 3
Neutrophil count decreased (Investigations) | 4 | 6
Platelet count decreased (Investigations) | 1 | 4
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 4 | 6
Anorexia (Metabolism and nutrition disorders) | 11 | 14
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 14
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 6
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 4
Hyponatremia (Metabolism and nutrition disorders) | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 7 | 15
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 4
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 7 | 8
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Nail loss (Skin and subcutaneous tissue disorders) | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No